CLINICAL TRIAL: NCT00607789
Title: A 12-Week, Double-Blind, Placebo-Controlled, Trial of Duloxetine Versus Placebo in the Treatment of Binge Eating Disorder and Comorbid Depressive Disorder.
Brief Title: Study of Duloxetine vs Placebo in Treatment of Binge Eating Disorder With Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Erik Nelson, Erik B. Nelson, MD & Susan McElroy, University of Cincinnati & Lindner Center of HOPE, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Nelson #2
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2012-11-14 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2012-09

CONDITIONS: Binge Eating; Depression
MeSH Terms: conditions — Bulimia; Depression | interventions — Duloxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duloxetine Group (Experimental): Start with 30 mg duloxetine hydrochloride capsule/day to be increased up to 120 mg per day.
  Interventions: Drug: Duloxetine
- Placebo Group (Placebo Comparator): Sugar pill with matching dosage as Duloxetine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 30 mg/day - 120 mg/day
  Other Names: Cymbalta
  Arms: Duloxetine Group
Drug: Placebo — identical to study drug
  Other Names: Sugar pill
  Arms: Placebo Group

SUMMARY:
The purpose of this research study is to test the safety of duloxetine and see what effects (good and bad) it has on the subject's binge eating disorder and comorbid depressive disorder (depression occurring with binge eating disorder) compared to placebo (inactive pill).

DETAILED DESCRIPTION:
This is a 12-week, double blind, randomized, placebo-controlled, parallel-group, flexible-dose study of duloxetine 60-120 mg/day in patients with BED and comorbid depressive disorders. Patients will be randomly assigned to either duloxetine 30 mg capsules or matching placebo at the baseline visit. The initial dose of study medication will be one 30 mg duloxetine capsule/day or placebo with a planned increase to 60 mg/day (2 X 30 mg) or matching placebo at the end of week 1. Further dose increases of 30 mg up to 120 mg/day will be allowed after the end of week two based on the investigators' assessment of efficacy and tolerability. Dosing will be either once per day or twice a day depending on tolerability. Patient visits will occur at screening and baseline and at the end of weeks 1, 2, 4, 6, 8, 10, and 12. Study drug will be tapered by 30 mg every 3 days at the end of the study.

ELIGIBILITY:
Inclusion criteria:

* Subjects must provide written informed consent of their own free will.
* Male or female outpatients.
* Age 18-65 years, inclusive.
* Subject must meet the DSM-IV criteria for a diagnosis of a depressive disorder (major depression, dysthymia, minor depression, or brief recurrent depression) for a duration of at least 1 month preceding and during the screening period.
* Subjects must meet the DSM-IV criteria for a diagnosis of binge eating disorder (BED) for at least the last 6 months. The DSM-IV criteria are as follows:

  1. Recurrent episodes of binge eating.
  2. The binge eating episodes are associated with at least three of the following: eating much more rapidly than normal; eating until uncomfortably full; eating large amounts of food when not feeling physically hungry; eating alone because of being embarrassed by how much one is eating; feeling disgusted with oneself, depressed, or feeling very guilty after overeating.
  3. Marked distress regarding binge eating.
  4. The binge eating occurs, on average, at least two days a week for the past six months.
  5. The episodes of binge eating do not occur exclusively during the course of bulimia nervosa or anorexia nervosa.
* Subjects will have an IDS score of at least 25 at the baseline visit.

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or of childbearing potential who are not using a medically acceptable, effective method of birth control. Women of childbearing potential include all pre-menopausal women biologically capable of becoming pregnant or contributing a fertilizable ovum. Medically acceptable methods of birth control include oral contraceptives, an intrauterine device, use of two combined barrier methods, or surgical sterilization.
* Patients who display significant risk for suicide.
* Patients who have received psychotherapy or behavioral therapy from a mental health professional as a part of previous treatment for MDD or obesity for at least 3 months prior to randomization.
* A DSM-IV diagnosis of alcohol or substance abuse or dependence, bulimia nervosa, or anorexia nervosa within the 6 months prior to randomization.
* Patients with a lifetime DSM-IV history of a psychotic disorder, a bipolar disorder, or dementia.
* Patients with a history of psychosurgery
* Patients with an Axis II disorder (personality disorders such as schizotypal, borderline, or antisocial), which might interfere with a diagnostic assessment, treatment, or compliance.
* Patients with clinically unstable medical disease.
* Patients with hepatic insufficiency
* Patients with end-stage renal disease or severe renal impairment
* Patients with a history of seizures, including febrile seizures in childhood.
* Patients requiring treatment with any drug which might interact adversely with or obscure the action of the study medication.
* Patients with a known hypersensitivity to duloxetine or any of the inactive ingredients of duloxetine (Cymbalta).
* Patients with uncontrolled narrow-angle glaucoma.
* Patients with clinically relevant abnormal laboratory results, specifically including hypokalemia.
* Patients who have received monoamine oxidase inhibitors, tricyclics, antipsychotics, lithium, or fluoxetine within four weeks prior to randomization.
* Patients who have received other psychoactive medications (including appetite suppressants) or any anti-obesity medications within one week prior to randomization.
* Patients who have received investigational medications or depot neuroleptics within three months prior to randomization.
* Patients previously enrolled in this study or who have previously been treated with duloxetine.
* Subject considered by the investigator as unable to be followed up throughout the entire duration of the study.
* Patients taking medications that inhibit the P450-2D6 hepatic isoenzyme

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik B Nelson, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati and Lindner Center of HOPE, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at the Lindner Center of HOPE location.
Pre-assignment Details: 64 participants were consented. 24 were not randomised: 21 did not meet entry criteria and 3 withdrew consent.
Groups:
- Duloxetine Group: 30-120 mg/day of duloxetine during a 12-week period
- Placebo Group: Placebo tablets (identical to duloxetine tablets), 30-120 mg/d given over 12-week period
Period: Overall Study
Arm/Group | Duloxetine Group | Placebo Group
Started | 20 (20 participants were randomized in each group) | 20
Completed | 13 | 14
Not Completed | 7 | 6
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Inadequate adherence | 3 | 0
Not completed — Lost to Follow-up | 0 | 5
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Duloxetine Group: Participants were randomized to 30-120 mg/day of duloxetine for 12 weeks
- Placebo Group: Participants who were randomized to 30-120 mg/day of sugar pill for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Duloxetine Group | Placebo Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.1) | 35.7 (10.4) | 40.05 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Binge Eating Days
Description: The mean number of binge days (days when the participant had one or more binge eating episodes) per week in the interval between visits (total number of binge days in the interval divided by number of days in the interval, then multiplied by 7).
Time Frame: 12 weeks
Population: The primary efficacy analysis was a longitudinal analysis comparing the rate of change of binge day frequency during the treatment period between groups.
Measure: Mean (Standard Deviation); unit: Mean Number of days
Groups:
- Duloxetine Group: Participants randomized to 30-120 mg/day of duloxetine for 12 weeks
- Placebo Group: Participants randomized to 30-120 mg/day of sugar pill for 12 weeks
Arm/Group | Duloxetine Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Mean Number of days | 4.3 (1.7) | 3.8 (1.7)
Statistical Analysis 1: Comparison: Duloxetine Group vs Placebo Group; The primary efficacy analysis was a longitudinal analysis comparing the rate of change of binge day frequency during the treatment period between groups. The same analysis was applied to binge episode frequency, weight, BMI, and scores on the CGI-Severity, YBOCS-BE, and IDS scales. The difference in rate of change was estimated by random regression methods; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 4.3, Standard Deviation 1.7

2. Secondary Outcome: Weekly Episodes
Description: The weekly frequency of binge episodes after baseline (number of binge eating days during the 12-week period divided by 7)
Time Frame: 12 weeks
Population: The secondary efficacy analysis was a longitudinal analysis comparing the rate of change of binge weeks frequency during the treatment period between groups.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Duloxetine Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Days | 4.7 (1.9) | 4.2 (2.6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The most frequent adverse events were: constipation, dry mouth, hyperhydrosis, and nausea.
Arm/Group | Duloxetine Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 20/20 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine Group (N=20) | Placebo Group (N=20)
Gastrointestinal problems (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant required a 48-hour hospitalization; the participant recovered fully and the event was thought not to be due to duloxetine.
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant who experienced gastrointestinal problems also had a sinus infection.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine Group (N=20) | Placebo Group (N=20)
Nausea (Gastrointestinal disorders) | 9 (9) | 3 (3)
Dry Mouth (General disorders) | 7 (7) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1)
Hyperhydrosis (Endocrine disorders) | 5 (5) | 2 (2) — Excessive sweating

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All trial data will be posted & published by the Lindner Center of HOPE (PI: Dr. Susan McElroy)